CLINICAL TRIAL: NCT05457621
Title: Evaluation of the Effectiveness and Tolerance of Effaclar Ultra Concentrated Serum in Women With Mandibular Acne for 3 Months (Including 2 Months of Treatment)
Brief Title: Effectiveness and Tolerance of Effaclar Serum in Women With Mandibular Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LRP19011-EFFACLAR SERUM
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Acne Vulgaris
Keywords: tri-acid complex serum; mandibular acne; microcomedones; maintenance regimen
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Participants attend 7 visits (screening visit, inclusion visit, 4 intermediate visits, final visit) and make a visit by phone call at Day48 hours. They apply the investigational product once daily (evening) for 2 months on the whole face and the accompanying product twice daily for 3 months on the whole face.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effaclar serum (Experimental): Participants are asked to apply Effaclar serum once daily in the evening on the whole face avoiding contact with eyes for 2 months.
  Interventions: Other: Effaclar serum

INTERVENTIONS:
Other: Effaclar serum — Effaclar serum has been formulated with an ultra-concentrated tri-acids complex for a synergetic action on skin and reinforced with soothing niacinamide for optimal tolerance. It acts in particular on imperfections and persistent marks due to acne.

SUMMARY:
The role of "dermocosmetics" in acne management is increasingly important, as many patients and even physicians now resort to them as first-line management in mild-to-moderate acne.

The aim of the study is to demonstrate the efficacy of the tested product on the appearance of acne lesions in 30 adult women suffering from acne in the mandible following an active anti-acne therapy (systemic or topical). This study includes 2 months of cosmetic treatment with EFFACLAR Ultra Concentrated Serum and one month of followup without any treatment but a moisturizer with a daily UV protection.

The investigational product has been formulated with an ultra-concentrated tri-acids complex for a synergetic action on skin and reinforced with soothing niacinamide for optimal tolerance.

This product is expected:

* to leave the skin clean and smooth,
* to help unblock pores,
* to exfoliate dead skin cells and help the skin to appear smoother, softer and pore-less,
* to be non-comedogenic.

DETAILED DESCRIPTION:
The study is performed in the Centre de Pharmacologie Clinique Appliqué à la Dermatologie (CPCAD), authorized by the French Regional Agency of Health (ARS) to perform biomedical research (Site agreement n°: 2016-04).

This clinical trial protocol and all amendments will be reviewed and approved by an appropriate Independent Ethics Committee (IEC) (Comité de Protection des Personnes (CPP)) located in France. The clinical trial cannot start before CPP approval.

The clinical trial is conducted under the sponsorship of Sponsor in compliance with the applicable international and local regulatory requirements as well as applicable International Council on Harmonisation (ICH) guidelines and in accordance with the Standard Operating Procedures (SOPs) for clinical trial conduct and monitoring from the assigned monitor.

All statistical tests will be two-sided and at the 5% level of significance. Normality tests will be at the 1% level of significance (Shapiro-Wilk).

Regarding the analysis of efficacy endpoints, quantitative parameters are analyzed using a linear mixed model for repeated measurements with Baseline and Time as fixed effects and Subject as random effect. Each time-point is compared to Baseline using a Dunes adjustment for multiplicity correction. For each fitted model, residual plots will be used to check the model assumptions. If there is an obvious deviation to these assumptions, the analysis is done on the rank-transformed data. Ordinal parameters (GEA) are analyzed using a cumulative link mixed model for repeated measurements with Baseline and Time as fixed effects and Subject as random effect. Each time-point will be compared to Baseline using a Dunnett adjustment for multiplicity correction.

The analysis of cosmeticity/acceptability questionnaire is descriptive only and for the analysis of safety endpoints, no statistical analysis is performed on safety. The data are presented descriptively.

As for the sample size determination, a total of 30 subjects completing the whole study allows to answer to the study objectives.

Clinical Research Associates (CRAs) and other applicable personnel are trained prior to study initiation to familiarize CRAs with the disease, the Standard Operating Procedures (SOP), the protocol and other study specific items.

Regarding the data management, the study data will be collected on an electronic data capture (EDC) set up by the Contract Research Organization (CRO). Computerized edit checks and review processes will be performed on an ongoing basis until all data clarifications are resolved. The data will be exported from a special database to be stored in appropriate format. After all data clarifications are resolved, coding is approved, and subject's evaluability is determined, the database will be locked.

ELIGIBILITY:
Inclusion Criteria:

* female subjects aged 20 years or above
* phototype II to IV
* mandibular acne (with or without diffuse acne)
* at baseline (Day0) a AFAST (Adult Female Acne Scoring Tool) score of 1 or 2 in the mandibular area and not over
* 15 non-inflammatory lesions and 5 inflammatory lesions minimum (screening and baseline)
* microcomedones on the mandibular area (visible with Vivacube measurement),

Exclusion Criteria:

* men
* female subject pregnant or lactating or who intends to conceive a child during the clinical trial or within one month after the last clinical trial visit
* facial acne without mandibular acne
* still undergoing medical treatment for acne at baseline (D0)
* intensively exposed to UV within the month preceding the baseline visit
* history of any severe disease or current condition (based on subject's interview and/or results of screening physical examination) which, in the opinion of the Investigator would put the subject at risk by participating in the study or would interfere significantly with the evaluation of study results (e.g. cancer, immune disorders)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Demonstrate the efficacy of Effaclar Ultra Concentrated Serum on the appearance of acne lesions in 30 adult women suffering from acne in the mandible following an active anti-acne therapy (systemic or topical).
Enrollment: 30 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
change in GEA (Global Evaluation Acne) score | from baseline to Day84
  evaluation of the acne grade by the investigator on a 6-point scale (from 0 Clear. No lesions to 5 Very severe)
change in Adult Female Acne Scoring Tool (AFAST) score | from baseline to Day84
  evaluation of the acne grade by the investigator on a 4-point scale
change in acne count | from baseline to Day84
  lesion count by the investigator: inflammatory lesions (papules, pustules, nodules) and non-inflammatory lesions (opened/closed comedones) on full face
change in the seborrhea evaluation | from baseline to Day84
  assessment performed by the investigator by visual inspection (gloss and shine aspect), and recorded using a 0-3 grading scale

SECONDARY OUTCOMES:
change in subject's and Investigator's global assessment of efficacy | from Day7 to Day84
  opinion given on the global efficacy of the study treatment at each visit (except Day0), using a 7-point scale
change in the quantity of sebum | from baseline to Day84
  evaluation, with a Sebumeter, of the quantity of sebum excreted to the skin surface. Measurements will be done about 12 h after the last application of any product and 3 h minimum after the last washing of the skin at controlled room temperature (21-25 °C).
change in the quality of life | Day0, Day14, Day28, Day56, Day84
  Cardiff Acne Disability Index (CADI) questionnaire with 5 questions
change in the global tolerance | from Day7 to Day84
  evaluation of the tolerance both by the investigator and the patient on a 5-point scale (from 0 None to 4 Very severe)
change in the sensitivity assessment by the investigator | from Day48 hours (phone call) to Day84
  assessment of the following signs: erythema, dryness, desquamation by the investigator on a 0-3 score
change in the sensitivity assessment by the participant | from Day48 hours (phone call) to Day84
  assessment of the following symptoms: itching, tingling, burning sensation by the patient on a 0-3 score

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Queille-Roussel, Study Director — Centre de Pharmacologie Clinique Applique a la Dermatologie
Locations (1):
- Centre de Pharmacologie Clinique Appliquée à la Dermatologie (CPCAD), Nice, France